CLINICAL TRIAL: NCT06338800
Title: One Session Virtual Reality During Ongoing Treatment for Anxiety: Feasibility in Children and Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Accare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSY-2324-S-0134
Record Dates: First submitted 2024-03-19; First posted 2024-04-01 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Disorders; Exposure; Social Anxiety Disorder
Keywords: Children; Adolescents; Virtual Reality Exposure; Anxiety disorders
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social

STUDY DESIGN:
Intervention Model Description: During ongoing treatment for their anxiety disorder 30 children and adolescents (8-18 years) with an anxiety disorder will receive a session of exposure with VR. Before the session expectations of VR exposure will be assessed. Before and after the session willingness to participate in exposure in vivo will be measured. During the session anxiety, idiosyncratic expectations, and self-efficacy are measured. After the session, positive effects, experiences, and negative side effects will be asked for.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One session VR Exposure (Experimental): All participants will receive one session exposure therapy with virtual reality during ongoing treatment.
  Interventions: Behavioral: One session exposure with Virtual Reality

INTERVENTIONS:
Behavioral: One session exposure with Virtual Reality — Participants will receive one session exposure with virtual reality from their therapists.

SUMMARY:
The goal of this study is to evaluate one session with exposure with Virtual Reality (VR) in in children and adolescents, aged 8-18 years with an anxiety disorder. The main questions it aims to answer are:

1. What are the expectations of children and adolescents and therapists with VR exposure?
2. What is the acceptability of the VR session (positive and negative effects)?
3. What are possible working mechanisms of VR exposure? During ongoing treatment, participants will receive a session of exposure with VR.

DETAILED DESCRIPTION:
Cognitive behavioral therapy is an effective treatment for anxiety disorders, with exposure as the most important working ingredient. Exposure therapy can be challenging to implement in face-to-face settings. Virtual reality (VR) has emerged as a promising tool for delivering exposure therapy.

In the current study, the researchers will examine children and adolescents that will participate in a single session of VR exposure during their regular treatment (n=30). Willingness to participate in exposure in vivo will be assessed directly before and directly after the session. During the session anxiety, idiosyncratic expectations, and self-efficacy will be assessed. Expectations will be measured before the session and acceptability after the session.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents 8-18 years old.
* Meeting Diagnostic and Statistical Manual of Mental Disorders -5 criteria for an anxiety disorder, based on a semi-structured interview (SCID-5 Jr, specific section) or clinical judgment of an experienced and authorized clinician.

Exclusion Criteria:

* Severe psychiatric symptoms other than anxiety disorder interfering with safety or warranting immediate intervention, e.g. psychosis or acute suicidality.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Willingness to participate in exposure in vivo | Directly before and immediately after the session
  Participants will be asked about their willingness to participate in exposure in vivo

SECONDARY OUTCOMES:
Idiosyncratic expectations | During the session
  Specific idiosyncratic expectations of the children and the adolescents, rated on a likert scale ranging from 0-10 (a higher score is a stronger belief).
Anxiety | During the session
  Anxiety of the children and adolescents will be rated on a likert-scale, subjective units of distress (SUD-scores) ranging from 0-10 (a higher score is more anxiety).
Expectations of Virtual Reality | Directly before the session
  Expectations of the session with virtual reality will be assessed with the Credibility and Expectancy Questionnaire for therapists and children.
Acceptability | Immediately after the session
  Acceptability of virtual reality exposure will be assessed with a questionnaire specifically designed for this study. Youth will be asked about positive and negative effects and their experiences.

IPD SHARING:
Plan to Share IPD: Yes
We will ask permission to share the data for potential future reanalysis, such as in a individual participant meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be requested after publication.